CLINICAL TRIAL: NCT02437305
Title: Melanoma Perception and Health Literacy in People of Color: A Targeted Educational Intervention
Brief Title: Melanoma Perception and Health Literacy in People of Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Roopal Kundu, Associate Professor in Dermatology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU00200459
Record Dates: First submitted 2015-04-16; First posted 2015-05-07 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2016-11

CONDITIONS: Melanoma
Keywords: Melanoma; People of Color
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABCDEs of Melanoma Skin Cancer (Experimental): A modified melanoma educational intervention that uses the "ABCDEs of Melanoma" pamphlet from the Skin Cancer Foundation but also incorporates the nomenclature "melanoma skin cancer"; indicates that melanoma is relevant for everyone regardless of race and ethnicity; includes images of melanoma on ethnic skin; informs people of the likelihood of melanoma developing in acral, subungual and mucosal surfaces; and provides guidance on self-skin examinations.
  Interventions: Behavioral: ABCDEs of Melanoma Skin Cancer
- ABCDEs of Melanoma (Active Comparator): A conventional melanoma educational intervention using the "ABCDEs of Melanoma" pamphlet from the Skin Cancer Foundation.
  Interventions: Behavioral: ABCDEs of Melanoma

INTERVENTIONS:
Behavioral: ABCDEs of Melanoma Skin Cancer — Modified melanoma educational intervention that is targeted towards people of color.
  Arms: ABCDEs of Melanoma Skin Cancer
Behavioral: ABCDEs of Melanoma — Conventional melanoma educational intervention.
  Arms: ABCDEs of Melanoma

SUMMARY:
This study will examine the effectiveness of a targeted, health literate educational intervention for people of color compared to a standard melanoma education pamphlet for increasing knowledge and promoting early melanoma detection. It is hypothesized that people of color are less aware of their risk for developing melanoma and that a targeted educational intervention will help increase knowledge and promote early melanoma detection especially in individuals with low health literacy.

DETAILED DESCRIPTION:
This targeted educational intervention will compare a standard melanoma education pamphlet with one that has been modified to target people of color. Both pamphlets will include the ABCDEs of melanoma, risk factors, prevention and treatment. In addition, the targeted pamphlet will incorporate the recommendations made by people of color in previous studies. The pamphlets will be randomized to subjects at a study visit along with a health literacy test and a questionnaire aimed at determining subjects' baseline melanoma knowledge and current melanoma prevention practices. 2 months post-intervention, a follow-up phone call will be made to assess subject knowledge retention and behavior change.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Self-identifies with one of the following races/ethnicities: African American, Asian/Pacific Islander, American Indian and Alaskan Native, or Hispanic

Exclusion Criteria:

* Not proficient in English
* Unable to give informed consent
* Does not self-identify with the following races/ethnicities: African American, Asian/Pacific Islander, American Indian and Alaskan Native, or Hispanic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roopal V Kundu, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Agbai ON, Buster K, Sanchez M, Hernandez C, Kundu RV, Chiu M, Roberts WE, Draelos ZD, Bhushan R, Taylor SC, Lim HW. Skin cancer and photoprotection in people of color: a review and recommendations for physicians and the public. J Am Acad Dermatol. 2014 Apr;70(4):748-762. doi: 10.1016/j.jaad.2013.11.038. Epub 2014 Jan 28. PMID 24485530
- [Background] Cormier JN, Xing Y, Ding M, Lee JE, Mansfield PF, Gershenwald JE, Ross MI, Du XL. Ethnic differences among patients with cutaneous melanoma. Arch Intern Med. 2006 Sep 25;166(17):1907-14. doi: 10.1001/archinte.166.17.1907. PMID 17000949
- [Background] Freeman HP. Poverty, culture, and social injustice: determinants of cancer disparities. CA Cancer J Clin. 2004 Mar-Apr;54(2):72-7. doi: 10.3322/canjclin.54.2.72. No abstract available. PMID 15061597
- [Background] Kundu RV, Kamaria M, Ortiz S, West DP, Rademaker AW, Robinson JK. Effectiveness of a knowledge-based intervention for melanoma among those with ethnic skin. J Am Acad Dermatol. 2010 May;62(5):777-84. doi: 10.1016/j.jaad.2009.08.047. Epub 2010 Mar 9. PMID 20219266
- [Background] Robinson JK, Joshi KM, Ortiz S, Kundu RV. Melanoma knowledge, perception, and awareness in ethnic minorities in Chicago: recommendations regarding education. Psychooncology. 2011 Mar;20(3):313-20. doi: 10.1002/pon.1736. PMID 20878831
- [Derived] Chao LX, Patterson SSL, Rademaker AW, Liu D, Kundu RV. Melanoma Perception in People of Color: A Targeted Educational Intervention. Am J Clin Dermatol. 2017 Jun;18(3):419-427. doi: 10.1007/s40257-016-0244-y. PMID 28035649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were consecutive patients seen for care at Northwestern Medicine's dermatology clinic in Chicago, IL between May and July 2015.
Period: Overall Study
Arm/Group | ABCDEs of Melanoma Skin Cancer | ABCDEs of Melanoma
Started | 50 | 50
Completed | 32 | 38
Not Completed | 18 | 12
Not completed — Lost to Follow-up | 18 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABCDEs of Melanoma Skin Cancer | ABCDEs of Melanoma | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Number; unit: participants]
  18-25 | 3 | 5 | 8
  26-50 | 26 | 29 | 55
  51-75 | 21 | 14 | 35
  76+ | 0 | 2 | 2
Gender [Count of Participants; unit: Participants]
  Female | 42 | 43 | 85
  Male | 8 | 7 | 15
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 39 | 39 | 78
  Asian/Pacific Islander | 5 | 6 | 11
  American Indian and Alaskan Native | 0 | 0 | 0
  Hispanic | 6 | 5 | 11
Education [Number; unit: participants]
  <12 years | 1 | 1 | 2
  High school | 2 | 4 | 6
  Some college/technical school | 12 | 11 | 23
  College graduate | 14 | 17 | 31
  Graduate/professional | 21 | 17 | 38
Personal history of skin cancer [Number; unit: participants]
  Yes | 1 | 1 | 2
  No | 49 | 49 | 98
Family history of skin cancer [Number; unit: participants]
  Yes | 1 | 6 | 7
  No | 49 | 44 | 93
Skin reaction to the sun [Number; unit: participants]
  Always burn/never tan | 3 | 1 | 4
  Usually burn/rarely tan | 3 | 1 | 4
  Rarely burn/usually tan | 18 | 24 | 42
  Never burn/always tan | 17 | 19 | 36
  None of these | 9 | 5 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Performed Regular Self-Skin Examinations
Description: The subject will complete 3 questionnaires: one pre-intervention, one immediately post-intervention and one 2 months post-intervention. 5 questions will assess whether or not the patient has completed skin-self examinations and knows which areas of the skin to pay attention to. The pre-intervention and 2 month post-intervention questionnaire will be evaluated to determine the number of participants that performed regular self-skin examinations.
Time Frame: 2 months post-intervention
Measure: Number; unit: participants
Arm/Group | ABCDEs of Melanoma Skin Cancer | ABCDEs of Melanoma
Number analyzed (Participants) | 32 | 38
participants
  Pre-I: perform skin self-exam | 8 | 16
  2MF: performed skin self-exam | 23 | 25
Statistical Analysis 1: Comparison: ABCDEs of Melanoma Skin Cancer vs ABCDEs of Melanoma; Test type: Superiority or Other; p = 0.048, McNemar — P-value compares the increase in skin self-exams from pre-intervention to 2-months follow-up between the 2 groups

2. Primary Outcome: Number of Participants With Correct Answers on Melanoma Perception Pre-intervention and 2 Months Post-intervention
Description: The subject will complete 3 questionnaires: one pre-intervention, one post-intervention, and one 2 months post-intervention. Several questions will assess the participants knowledge of general melanoma, what it looks like and what are its risk factors. To determine participant retention, the pre-intervention and 2 month post-intervention questionnaires will be evaluated.
Time Frame: 2 months post-intervention
Measure: Number; unit: participants
Arm/Group | ABCDEs of Melanoma Skin Cancer | ABCDEs of Melanoma
Number analyzed (Participants) | 32 | 38
participants
  Pre-I: Melanoma is a type of skin cancer | 27 | 28
  2MF: Melanoma is a type of skin cancer | 31 | 36
  Pre-I: Sun exposure is linked to melanoma | 23 | 29
  2MF: Sun exposure is linked to melanoma | 30 | 36
  Pre-I: Knows the warning signs of melanoma | 24 | 23
  2MF: Knows the warning signs of melanoma | 30 | 33
Statistical Analysis 1: Comparison: ABCDEs of Melanoma Skin Cancer vs ABCDEs of Melanoma; Test type: Superiority or Other; p > 0.50, McNemar — P-value compares the increase in knowledge from pre-intervention to 2-months follow-up between the 2 groups

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | ABCDEs of Melanoma Skin Cancer | ABCDEs of Melanoma
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
Small sample size and high dropout rate; recruitment from dermatology clinic patients with a majority having college degrees or higher so the study results are less generalizable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No